CLINICAL TRIAL: NCT04270032
Title: To Build and Evaluate a Precise Diagnosis, Therapy Assessment and Prognosis Prediction Model of Breast Cancer Based on Artificial Intelligence
Brief Title: Using Deep Learning Methods to Analyze Automated Breast Ultrasound and Hand-held Ultrasound Images, to Establish a Diagnosis, Therapy Assessment and Prognosis Prediction Model of Breast Cancer.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of the Fourth Military Medical University (Other)
Collaborators: Seoul National University Bundang Hospital (Other); Xidian University (Other); Shenzhen University (Other)
Responsible Party: Principal Investigator, Song Hongping, Principal Investigator, The First Affiliated Hospital of the Fourth Military Medical University
Other Study IDs: AI-Breast-US
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- malignant group: women with malignant lesions confirmed by pathology
  Interventions: Diagnostic Test: ABUS and HHUS
- benign group: women with benign lesions confirmed by pathology or stable in follow-up > 2 years
  Interventions: Diagnostic Test: ABUS and HHUS
- normal group: women have normal images with follow up > 2 years
  Interventions: Diagnostic Test: ABUS and HHUS

INTERVENTIONS:
Diagnostic Test: ABUS and HHUS — Using deep learning method to analyze and extract the features of automated breast ultrasound and hand-held ultrasound images

SUMMARY:
The purpose of this study is using a deep learning method to analyze the automated breast ultrasound (ABUS) and hand-held ultrasound(HHUS) images, establish and evaluate a diagnosis, therapy assessment and prognosis prediction model of breast cancer. The model would provide important references for further early prevention, early diagnosis and personalized treatment.

DETAILED DESCRIPTION:
1. Establishing a database By collecting ABUS, HHUS and comprehensive breast images data, essential information, clinical treatment information, prognosis, and curative effect information, a complete breast image database is constructed.
2. Marking ABUS images Three doctors use a semi-automatic method to frame the lesions on the image.
3. Building the model Using the deep learning method to preprocess, analyze and train the marked images, and finally get a model diagnosis, efficacy evaluation and prognosis prediction model of breast cancer.
4. Evaluating the model 1）Self-validation： Analyze the sensitivity, AUC of the breast cancer diagnosis model and the false-positive number on each ABUS volume.

2) Compared the sensitivity, AUC and the false-positive number with a commercial diagnosis model.

3)To test the screening and diagnostic efficacy of computer-aided diagnosis systems through prospective or retrospective studies.

4)By analyzing the size and characteristics of the lesions after neoadjuvant chemotherapy, and predicting the OS and DFS time, the therapy assessment and prognosis prediction model were evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients over 18 years old who come to the two centers for physical examination or treatment;
2. Complete basic information and image data

Exclusion Criteria:

1. There is no complete ABUS and HHUS images data;
2. The image quality is poor;
3. In multifocal breast cancer, the correlation between the tumor in the image and the postoperative pathological examination is uncertain.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female patients over 18 years old from two countries (China and Korea).
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
sensitivity | 4 years
  Proportion of corrected-marked malignant lesions by the model
false-positive per volume | 4 years
  the number of uncorrected-marked malignant lesions by the model
area under curve | 4 years
  area under receiver operating characteristic (ROC) curve in percentage (%)
overall survival(OS) time | up to 10 years
  It measures the time from the date of cancer diagnosis to any cause of death.
Disease-free survival (DFS) time | up to 5 years
  The time that the patient is free of the signs and symptoms of a disease after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hongping Song, MD, Principal Investigator — Xijing hospital of The fourth military medical university
Locations (1):
- The First Affiliated Hospital of Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided